CLINICAL TRIAL: NCT00724165
Title: Seamos Activas: Increasing Physical Activity Among Latinas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Dr.Bess Marcus, Professor and Chair, Department of Family and Preventive Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: R21NR009864 (NIH); R21NR009864 (NIH)
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Inactivity
Keywords: physical activity; Latinas
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Intervention
- 2 (Active Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention — Culturally-modified, individually tailored physical activity print materials
  Arms: 1
Behavioral: Control — Bilingual health education booklets
  Arms: 2

SUMMARY:
The overarching goal of this project is to develop a culturally congruent intervention to increase levels of physical activity among sedentary Latinas (i.e., Latina/Hispanic women). The first phase will involve culturally and linguistically modifying an existing evidenced-based intervention, founded on the Transtheoretical Model and Social Cognitive Theory, to target sedentary Latinas. Then, we will conduct a pilot randomized clinical trial to test whether the culturally-modified individually tailored intervention increases physical activity levels in comparison to standard care comprised of bilingual health education booklets.

DETAILED DESCRIPTION:
While the general United States population is suffering from an epidemic of sedentary lifestyle, Latinos are even more sedentary than their non-Hispanic white counterparts. Notably, Latinos suffer from greater rates of morbidity and mortality of conditions associated with being sedentary than non-Hispanic whites. One concern is that due to cultural artifacts, socioeconomic circumstances, and language barriers, Latinos have limited access to public health interventions that promote active lifestyles. The current study will advance nursing science by using a theory-based computer-run expert system to provide an effective physical activity intervention for this underserved population. The consent form was completed by all participants and describes the nature and purpose of the study, procedure, risks and benefits to participating, alternative therapies available, and confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary (i.e., participating in moderate or vigorous physical activity two days per week or less for 30 minutes or less each day) women ages 18 to 65 who self-identify as Latina (or of a group defined as Hispanic/Latino by the Census Bureau) are eligible for participation

Exclusion Criteria:

* Exclusion criteria are history of coronary heart disease (history of myocardial infarction or symptoms of angina), diabetes, stroke, osteoarthritis, osteoporosis, orthopedic problems, or any other serious medical condition that would make physical activity unsafe. Other exclusion criteria will include individuals who report consuming three or more alcoholic drinks per day, current or planned pregnancy, planning to move from the area within the next six months, current suicidal ideation or psychosis, current clinical depression, hospitalization due to a psychiatric disorder in the past 3 years, BMI above 40, and/or taking medication that may impair physical activity tolerance or performance (e.g., beta blockers). Participants in the pilot study must also agree to be assigned to one of the two intervention conditions.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2006-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Self-Reported physical activity | Baseline, 3 months, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bess H Marcus, PhD, Principal Investigator — Alpert Medical School of Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Pekmezi DW, Neighbors CJ, Lee CS, Gans KM, Bock BC, Morrow KM, Marquez B, Dunsiger S, Marcus BH. A culturally adapted physical activity intervention for Latinas: a randomized controlled trial. Am J Prev Med. 2009 Dec;37(6):495-500. doi: 10.1016/j.amepre.2009.08.023. PMID 19944914